CLINICAL TRIAL: NCT07036159
Title: A Phase 2a, Open Label, Randomized, Interventional Study to Assess the Safety and Immunogenicity of Alternative Vaccination Regimens and Reduced Antigen Doses of RTS,S/AS01E Vaccine in Healthy Children Aged 5-60 Months in a Malaria-endemic Area
Brief Title: A Study to Assess the Safety and Immunogenicity of a Vaccine Against Malaria in Healthy Children Aged 5-60 Months
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 223247; 2024-000563-20 (EudraCT Number)
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Malaria
Keywords: Parasitic disease; Plasmodium falciparum; Malaria; Safety; Immunogenicity; Healthy children
MeSH Terms: conditions — Malaria; Parasitic Diseases; Malaria, Falciparum | interventions — RTS,S-AS01E vaccine; RTS malaria vaccine

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Groups 1 to 3 (Experimental): Participants receive 3 doses of RTS,S/AS01E vaccine on Day 1, Month 1, and Month 2.
  Interventions: Biological: RTS,S/AS01E vaccine
- Groups 4 and 5 (Experimental): Participants receive 3 doses of RTS,S/AS01E vaccine on Day 1, Month 1, and Month 7.
  Interventions: Biological: RTS,S/AS01E vaccine
- Groups 6 and 7 (Experimental): Participants receive 3 doses of RTS,S/AS01E vaccine on Day 1, Month 2, and Month 7.
  Interventions: Biological: RTS,S/AS01E vaccine

INTERVENTIONS:
Biological: RTS,S/AS01E vaccine — RTS,S/AS01E vaccine will be administered intramuscularly.
  Other Names: Mosquirix

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of reduced antigen doses and alternative vaccination regimes for RTS,S/AS01E in healthy children aged 5-60 months in a malaria-endemic area.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants aged 5 to 60 months at the time of the first vaccination, who have previously completed the World Health Organization (WHO) Expanded Programme on Immunization (EPI) vaccinations or for younger infants have received all required vaccinations at point of recruitment according to the schedule for the country where the study is conducted.
2. Participants' parent(s)/Legally Acceptable Representative(s) (LAR), in the opinion of the investigator, can and will comply with the requirements of the protocol (eg, completion of the diaries, returning for follow-up visits).
3. Written or witnessed/thumb-printed informed consent obtained from the participant's parent(s)/LAR prior to performance of any study-specific procedure.
4. Healthy, as established by medical history and clinical examination.
5. Negative for human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV).
6. With hemoglobin levels >8 g/dL.
7. Born after a gestation period of ≥37 weeks.

Exclusion Criteria:

1. Progressive, unstable, or uncontrolled clinical conditions.
2. History (known or suspected) of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccine.
3. Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
4. Clinical conditions representing a contraindication to IM vaccination or blood draws.
5. Any behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the participant's ability to participate in the study.
6. Recurrent history of or uncontrolled neurological disorders or seizures.
7. Undernutrition, defined as WHO Z-score less than -2 standard deviation.
8. Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant as a result of participation in the study, for example, any major congenital defects.
9. Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by physical examination and medical history.
10. Administration of long-acting immune-modifying drugs (eg, infliximab) during the study period starting 3 months before the first dose of study vaccine or planned administration during the study period.
11. Prior receipt of a malaria vaccine (registered or experimental).
12. Use of any investigational or non-registered product (drug, vaccine, or medical device)* other than the study vaccine during the period starting 30 days before the first dose of study vaccine (Day -30 to Day 1), or planned use during the study period.

    *Use of herbs and traditional treatments is not considered an exclusion criterion.
13. Planned administration of a vaccine not foreseen by the study protocol or the country EPI in the period starting 14 days before each dose and ending 28 days after the last dose of study vaccine administration*, with the exception of flu vaccines and vaccines administered as part of a public health vaccination campaign*.

    *If emergency mass vaccination for an unforeseen public health threat (eg, a pandemic) is organized by public health authorities outside the routine immunization program, the time period described above can be reduced, provided the vaccination is used according to the local governmental recommendations and the Sponsor is notified.

    Under such circumstances, a participant may be considered eligible for study enrollment and/or study vaccine administration after the appropriate window for delay has passed, if the participant is confirmed to be eligible after inclusion/exclusion criteria have been re checked.
14. Administration of immunoglobulins and/or any blood products or plasma derivatives, or bone marrow transplantation, during the period starting 3 months before the first dose of study vaccine or planned administration during the study period.
15. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first vaccine dose or planned administration during the study period. For corticosteroids, this means prednisone ≥0.5 mg/kg/day or 20 mg/day, whichever is the maximum dose for pediatric participants. Inhaled and topical steroids are allowed.
16. Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug or invasive medical device).
17. Any study personnel's immediate dependents, family, or household members.
18. Child in care.

Ages: 5 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 238 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-04-23 (Estimated); Study Completion 2027-04-23 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Concentrations (GMCs) of anti-NANP immunoglobulin G (IgG) antibodies | 12 months post-Dose 3 (Month 14 for Groups 1 to 3 and Month 19 for Groups 4 and 5 and Groups 6 and 7)

SECONDARY OUTCOMES:
Area under the curve (AUC) of anti-NANP IgG antibodies | At Month 7 and 19
GMC of anti-NANP IgG antibodies | At Month 0, 1, 2, 3, 7, 8, 14, and 19
Number of participants with a greater than or equal to (>=) 2-fold and a (>=) 4-fold increase from pre-Dose 1 in IgG antibody concentration | At Month 0, 1, 2, 3, 7, 8, 14, and 19
Number of participants with solicited administration site events | Up to 7 days after each vaccine administration (vaccine administered on Day 1, Month 1, Month 2, and Month 7)
  Solicited administration site events include pain, redness, and swelling at administration site.
Number of participants with solicited systemic events | Up to 7 days after each vaccine administration (vaccine administered on Day 1, Month 1, Month 2, and Month 7)
  Solicited systemic events include fever, irritability/fussiness, loss of appetite, sleepiness/drowsiness, and vomiting.
Number of participants with unsolicited adverse events (AEs) | Within 30 days after each study vaccine administration (vaccine administered on Day 1, Month 1, Month 2, and Month 7)
  An unsolicited AE is an AE that is either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Number of participants with serious adverse events (SAEs) | From first study vaccine administration (Day 1) to the end of the study (Month 19)
  An SAE is defined as any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongs existing hospitalization, results in disability/incapacity, or other medically significant events.
Number of participants with SAEs | From first study vaccine administration (Day 1) to 12 months after the last study vaccine administration (Month 14 for Groups 1 to 3 and Month 19 for Groups 4 and 5 and Groups 6 and 7)
Number of participants with adverse events of special interest (AESIs) | Up to 7 days after each vaccine administration (vaccine administered on Day 1, Month 1, Month 2, and Month 7)
  AESIs include febrile convulsion that are defined as seizures that occur in febrile children between the ages of 6 and 60 months who do not have an intracranial infection, metabolic disturbance, or history of afebrile seizures.
Number of participants with AEs/SAEs leading to withdrawal from the study and/or discontinuation of study vaccine | From first study vaccine administration (Day 1) to the end of the study (Month 19)
GMC of anti-hepatitis B surface antigens (HBs) antibody concentrations (IgG) | At Month 0, 1, 2, 3, 7, 8, 14, and 19
Number of participants achieving anti-HBs IgG levels above 6.2 International Units per liter (IU/L) and 10.0 IU/L | At Month 0, 1, 2, 3, 7, 8, 14, and 19
Geometric mean fold increase over pre-Dose 1 for anti-HBs IgG | At Month 0, 1, 2, 3, 7, 8, 14, and 19

CONTACTS AND LOCATIONS:
Overall Officials: Julien M Nyombayire, MD, MSc, Principal Investigator — Center for Family Health Research; Mossi Nzeyimana, MD, Principal Investigator — Rinda Ubuzima Gatenga Medicalized Health Center University of Rwanda
Locations (1):
- GSK Investigational Site, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf